CLINICAL TRIAL: NCT02944552
Title: The Multi Center, Randomized, Double-blind, Positive Controlled Phase II Clinical Trial of Bicyclol Tablets in the Treatment of Acute Drug-induced Liver Injury
Brief Title: The Multi Center, Randomized, Double-blind, Positive Controlled Study of Bicyclol in the Treatment of Acute DILI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drug Induced Liver Disease Study Group (Other)
Collaborators: Beijing Union Pharmaceutical Factory Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YL-SHC-2015
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Drug-Induced Acute Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — bicyclol; polyene phosphatidylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose group (Experimental): Patients in the low dose group administrated bicyclol tablet 25mg orally, three times daily for 4-8 weeks.
  Interventions: Drug: bicyclol tablet 25mg
- high dose group (Experimental): Patients in the high dose group administrated bicyclol tablet 50mg orally, three times daily for 4-8 weeks.
  Interventions: Drug: bicyclol tablet 50mg
- positive drug control group (Active Comparator): Patients in the positive drug control group administrated polyene phosphatidylcholine capsule 456mg orally, three times daily for 4-8 weeks.
  Interventions: Drug: polyene phosphatidylcholine capsule 456mg

INTERVENTIONS:
Drug: bicyclol tablet 25mg — Patients in the low dose group administrated bicyclol tablet 25mg, one bicyclol blank analog tablet and two polyene phosphatidylcholine blank analog capsules orally, three times daily for 4-8 weeks.
  Other Names: bicyclol blank analog tablet; polyene phosphatidylcholine blank analog capsule
  Arms: low dose group
Drug: bicyclol tablet 50mg — Patients in the high dose group administrated bicyclol tablet 50mg and two polyene phosphatidylcholine blank analog capsules orally, three times daily for 4-8 weeks.
  Other Names: polyene phosphatidylcholine blank analog capsule
  Arms: high dose group
Drug: polyene phosphatidylcholine capsule 456mg — Patients in the positive drug control group administrated polyene phosphatidylcholine capsules 456mg and two bicyclol blank analog tablets orally, three times daily for 4-8 weeks.
  Other Names: bicyclol blank analog tablet
  Arms: positive drug control group

SUMMARY:
The study adopted the superiority design of multi center, randomized, double-blind, positive control drug, dose finding, using two simulation skills. The qualified subjects, according to the ratio of 1:1:1, were randomized into low dose group, high dose group and positive drug control group, and received a treatment course of 4-8 weeks, all individuals were followed up for 4 weeks after drug withdrawal.

DETAILED DESCRIPTION:
Explore the safety and efficacy of different doses of bicyclol in treatment of acute drug-induced liver injury using polyene phosphatidylcholine capsule as the positive control drug.

The study adopted the design of multi center, randomized, double-blind, dose finding, positive control drug, superiority test, using two simulation skills. The qualified subjects, according to the ratio of 1:1:1, were randomized into low dose group and high dose group and positive drug control group, and received a treatment course of 4-8 weeks, all individuals were followed up for 4 weeks after drug withdrawal.

ELIGIBILITY:
Inclusion criteria:

1. 18-75 years old, male or female;
2. Meet the standard of clinical diagnosis of acute drug-induced liver injury, the RUCAM causality scale score is more than or equal to 6 points. If the RUCAM causality scale score is 3-5,the subject needs three liver disease experts to confirm whether he is DILI patient, at least two of three liver disease experts should have the same judgment;
3. The serum ALT is between 3and 20 times ULN, but TBiL is less than or equal to 2 times ULN;
4. Liver biochemical indexes(ALT,AST,ALP,GGT,TBiL,albumin,prothrombin time) abnormalities lasted less than 90 days;
5. Patients can understand the nature of the experiment, the nature of the disease, the characteristic of drugs, related treatment methods and the risk they may need to bear if they participate in the test, and sign the informed consent.

Exclusion criteria:

1. Occurrent liver injury caused by other reasons, such as viral hepatitis, alcoholic liver disease, nonalcoholic fatty liver disease etc;
2. Acute liver failure or liver function decompensation patient perform, such as hepatic encephalopathy, ascites, albumin is less than or equal to 35g / L, The international standardized ratio (INR) of thrombin is more than 1.5;
3. Serum creatinine is more than 1.5 times ULN;
4. Severe or life-threatening heart, lung, brain, kidney, gastrointestinal and systemic diseases;
5. Taking drugs that may affect observation of curative effect of the experimental drug during the study;
6. Allergy or intolerance to experimental drugs;
7. With no ability to express their complaints, such as mental illness and severe neurosis patient;
8. The patient can not cooperate and poor compliance;
9. Pregnant and lactating women or women preparing for pregnancy;
10. The patient participated in other clinical trials in 3 months before entering this study;
11. Using other liver-protective drugs except ursodeoxycholic acid or ademetionine within three days;
12. The researchers believe not suitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The decline range of serum ALT after 4 weeks of treatment | after 4 weeks of treatment
  The decrease value of serum ALT after 4 weeks of treatment compared to the baseline

SECONDARY OUTCOMES:
The decrease value of serum AST compared to the baseline of treatment for 1, 2, 4, 6, 8 weeks and follow-up for 2, 4 weeks | after 1, 2, 4, 6, 8 weeks treatment and follow-up for 2, 4 weeks
  The decrease value of serum AST compared to the baseline
The decrease value of serum ALT compared to the baseline of treatment for 1, 2, 6, 8 weeks and follow-up for 2, 4 weeks | after 1, 2, 6, 8 weeks treatment and follow-up for 2, 4 weeks
  The decrease value of serum ALT compared to the baseline
The decrease rate of serum ALT compared to the baseline of treatment for 1, 2, 4, 6, 8 weeks and follow-up for 2, 4 weeks | after 1, 2, 4, 6, 8 weeks treatment and follow-up for 2, 4 weeks
  The decrease rate of serum ALT compared to the baseline
The time from treatment to ALT normalization | treatment period
  The time from treatment to ALT normalization
The ratio of subjects whose ALT and AST declined more than 50% compared to the base line of treatment for 1, 2, 4, 6, 8 weeks and follow-up for 2, 4 weeks | after 1, 2, 4, 6, 8 weeks treatment and follow-up for 2, 4 weeks
  The ratio of subjects whose ALT and AST declined more than 50% compared to the base line
The serum ALT and AST normalization rate of treatment for 1, 2, 4, 6, 8 weeks and follow-up for 2, 4 weeks | after 1, 2, 4, 6, 8 weeks treatment and follow-up for 2, 4 weeks
  The serum ALT and AST normalization rate
The area under curve of ALT and AST of treatment for 1, 2, 4, 6, 8 weeks and follow-up for 2, 4 weeks | after 1, 2, 4, 6, 8 weeks treatment and follow-up for 2, 4 weeks
  The area under curve of ALT and AST

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mao, Study Chair — RenJi Hospital; Chengwei Chen, Study Chair — No.85 hospital of PLA
Locations (17):
- China (17):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The second affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - The First affiliated Hospital of Xinxiang Medical University, Weihui, Henan
  - Henan Infectious Diseases Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Renji Hospital ，Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - No.85 hospital of PLA, Shanghai, Shanghai Municipality
  - Ruijin Hospital ，Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Tianjin Haihe Hospital, Tianjin, Tianjin Municipality
  - Shanghai Lung Hospital, Shanghai

REFERENCES:
- [Derived] Tang J, Gu J, Chu N, Chen Y, Wang Y, Xue D, Xie Q, Li L, Mei Z, Wang X, Li J, Chen J, Li Y, Yang C, Wang Y, Shang J, Xie W, Hu P, Li D, Zhao L, Lan P, Wang C, Chen C, Mao Y. Efficacy and safety of bicyclol for treating patients with idiosyncratic acute drug-induced liver injury: A multicenter, randomized, phase II trial. Liver Int. 2022 Aug;42(8):1803-1813. doi: 10.1111/liv.15290. Epub 2022 May 25. PMID 35567757